CLINICAL TRIAL: NCT04226924
Title: A Randomized, Double-Blind, Placebo-Controlled Efficacy and Safety Trial of Trehalose for the Treatment of
Brief Title: Treatment of Oculopharyngeal Muscular Dystrophy With Trehalose
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of funding for company
Sponsor: Bioblast Pharma Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BB-OPMD-202
Record Dates: First submitted 2019-07-15; First posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Oculopharyngeal Muscular Dystrophy
Keywords: OPMD; DMOP; Dysphagia
MeSH Terms: conditions — Muscular Dystrophy, Oculopharyngeal; Deglutition Disorders | interventions — Trehalose

STUDY DESIGN:
Intervention Model Description: The study includes a 24-week blinded treatment period during which patients will receive weekly infusions of trehalose or placebo, followed by a 24-week open-label extension period during which all patients will receive weekly infusions of trehalose.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The Treatment Period of the study is double-blind. The Extension Period is open label.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trehalose (Experimental): Trehalose 9% solution: The dose is 0.75 g/kg administered IV over 60 ± 5 minutes once weekly.
  Interventions: Drug: Trehalose
- 0.9% Normal Saline (Placebo Comparator): Normal saline: weight-based volume administered IV over 60 ± 5 minutes once weekly.
  Interventions: Drug: Trehalose

INTERVENTIONS:
Drug: Trehalose — 90 mg/ml trehalose solution for IV infusion

SUMMARY:
BB-OPMD-202 is a randomized, double-blind, placebo-controlled study of IV trehalose for treatment of OPMD. The study includes a 4-week screening period, a 24-week blinded treatment period during which patients will receive weekly infusions of trehalose or placebo, followed by a 24-week open-label extension period during which all patients will receive weekly infusions of trehalose. Patients will undergo a safety follow-up assessment 4 weeks after their last treatment.

DETAILED DESCRIPTION:
After signing informed consent, patients will undergo two rounds of ice-cold water and nectar drinking tests at least 1 week apart to confirm oropharyngeal dysfunction. Patients who have confirmed oropharyngeal dysfunction, i.e., an ice-cold water drinking test time of 8 seconds or greater at both rounds, in addition to an SSQ score of >235, will be enrolled. Baseline values for all safety and efficacy parameters will be established during the screening period. Patients will be randomized in a 1:1 ratio, to trehalose or placebo, at the time of enrollment. Randomization will be stratified according to the patient's score on the SSQ at screening (≤ 799 or ≥ 800).

Patients randomized to trehalose will receive a 1-hour IV infusion of trehalose at a dose of 0.75 g/kg weekly for 24 weeks. Patients randomized to placebo (normal saline) will receive a weight-based equal volume of placebo weekly for 24 weeks.

After Week 24, patients may transition to an open-label extension of the study (extension period). During the extension period, patients will be treated with weekly infusion of trehalose at a dose of 0.75 g/kg for 24 weeks, followed by a 4-week safety follow-up (total duration of study = 56 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Genetically confirmed OPMD with a (GCN)13 size PABPN1 mutation
* A score greater than 235 on the Sydney Swallow Questionnaire at screening
* Confirmation of oropharyngeal dysfunction by abnormal ice-cold water drinking test result, defined as drinking 80 cc of ice-cold water in ≥ 8 seconds at both drinking tests (at least 1 week apart) during the screening period

Exclusion Criteria:

* History of pharyngeal myotomy.
* Esophageal dilatation within the last 12 months.
* Treatment with botulinum toxin (any location) within 1 year prior to screening.
* Diagnosis of any other muscle disorder.
* Prior head and neck surgery or radiation.
* Oropharyngeal injury or oropharyngeal cancer.
* Other esophageal disease that may be the cause of the dysphagia.
* Previously diagnosed with diabetes or a hemoglobin A1c (HgbA1c) result > 6.0% at screening.
* Prior treatment with IV trehalose.
* Known hypersensitivity to trehalose.
* Non-ambulatory (Use of a cane or short leg braces are permitted).
* Prior history of stroke (ischemic or hemorrhagic).
* Pregnancy or breast feeding.
* History of alcohol or drug abuse within the last 5 years.
* Evidence of hepatitis B, hepatitis C, or HIV infection at screening.
* Currently receiving anti-coagulant treatment (e.g., warfarin, enoxaparin) other than anti-platelet treatments, which are not a reason for exclusion.
* Currently participating in another clinical trial or has completed an interventional trial less than 90 days prior to planned first dosing.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2018-02-15 (Estimated); Study Completion 2018-08-15 (Estimated)

PRIMARY OUTCOMES:
Drinking Test Time | 24 weeks
  Change from baseline in timed drinking tests with 80 cc of ice-cold water and nectar.

SECONDARY OUTCOMES:
Muscle Strength Testing | 24 weeks
  Change from baseline in strength tests in selected muscle groups as measured by a handheld dynamometer
Stair Climb Test | 24 weeks
  Change from baseline in functional muscle testing as measured by the Stair Climb test
Timed Up and Go Test | 24 weeks
  Change from baseline in functional muscle testing as measured by the Timed Up and Go (TUG) test
30-Second Lift Test | 24 weeks
  Change from baseline in functional muscle testing as measured by 30-Second Lift test
EuroQol-5D-5L | 24 weeks
  Change from baseline in health status using the EuroQol-5D-5L Questionnaire
Swallowing Quality of Life | 24 weeks
  Change from baseline in quality of life using modified Swallowing Quality of Life Questionnaire
Sydney Swallow Questionnaire | 24 weeks
  Change from baseline in quality of life using Sydney Swallow Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Brais, MD, Principal Investigator — McGill University
Locations (3):
- Canada (3):
  - Ecogene-21, Chicoutimi, Quebec
  - Montreal Neurological Institute and Hospital, Montreal, Quebec
  - CHU de Québec-Université Laval- Hôpital Enfant-Jésus, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No